CLINICAL TRIAL: NCT02598128
Title: Study to Evaluate Safety, Tolerability and Fat Absorption Using a Novel Enteral Feeding In-line Digestive Enzyme Cartridge (RELIZORB) in Patients With Cystic Fibrosis Receiving Enteral Feeding
Brief Title: Safety, Tolerability and Fat Absorption Using Enteral Feeding In-line Enzyme Cartridge (Relizorb)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcresta Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: ALCT-0000497
Record Dates: First submitted 2015-11-03; First posted 2015-11-05 (Estimated); Results first posted 2017-01-20 (Estimated); Last update posted 2017-01-25 (Estimated); Status verified 2017-01

CONDITIONS: Exocrine Pancreatic Insufficiency
MeSH Terms: conditions — Exocrine Pancreatic Insufficiency

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- RELiZORB (Experimental): Treatment (RELiZORB)
  Interventions: Device: RELiZORB
- Control (Placebo Comparator): Placebo control
  Interventions: Device: Placebo

INTERVENTIONS:
Device: RELiZORB — Peptamen 1.5 received Period A and Period B (washout only). Impact Peptide 1.5 received Period B (Days 1 and 9 only) and Period C.
  Other Names: Peptamen 1.5; Impact Peptide 1.5
  Arms: RELiZORB
Device: Placebo — Sham device
  Arms: Control

SUMMARY:
Protocol ALCT-0000497 is a multicenter safety, tolerability and fat absorption study that anticipates enrolling 35 male and female subjects (pediatric and adult) with cystic fibrosis. Subjects with confirmed exocrine pancreatic insufficiency will use a novel enteral feeding in-line digestive enzyme cartridge (RELiZORB) connected to enteral pump sets.

DETAILED DESCRIPTION:
Protocol ALCT-0000497 consists of three distinct study periods as follows:

1. In Period A (7 days), subjects will receive Peptamen 1.5 enteral feedings at home.
2. In Period B (11 days), subjects will be randomized to either Group A (active investigational then placebo control) or Group B (placebo control then active investigational) and receive Impact Peptide 1.5 on Days 1 and 9. During the 8-day washout period between Days 1 and 9, subjects will receive Peptamen 1.5.
3. In Period C (9 days), subjects will use RELiZORB during nocturnal enteral feedings with Impact Peptide 1.5.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed CF diagnosis with 2 clinical features
2. Documented history of EPI
3. Enteral formula use minimum of 4x/week
4. Written informed consent or assent, as applicable

Exclusion Criteria:

1. Uncontrolled diabetes mellitus
2. Signs and symptoms of liver cirrhosis or portal hypertension
3. Lung/liver transplant
4. Active cancer currently receiving cancer treatment
5. Crohn's or celiac disease, infectious gastroenteritis, sprue, lactose intolerant, inflammatory bowel disease
6. DIOS or fibrosing colonopathy

Ages: 4 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 34 (Actual)
Dates: Start 2015-11; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Russell G. Clayton, Sr., DO, Study Director — Chief Medical Officer, Alcresta Therapeutics, Inc.
Locations (11):
- United States (11):
  - Children's Hospital of Los Angeles, Los Angeles, California
  - St. Luke's Cystic Fibrosis Center of Idaho, Boise, Idaho
  - Riley Hospital for Children at Indiana University Health, Indianapolis, Indiana
  - Maine Medical Center, Portland, Maine
  - Children's Mercy Hospital, Kansas City, Missouri
  - Cardinal Glennon Children's Medical Center, St Louis, Missouri
  - Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Monroe Carell Junior Children's Hospital at Vanderbilt, Nashville, Tennessee
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Freedman S, Orenstein D, Black P, Brown P, McCoy K, Stevens J, Grujic D, Clayton R. Increased Fat Absorption From Enteral Formula Through an In-line Digestive Cartridge in Patients With Cystic Fibrosis. J Pediatr Gastroenterol Nutr. 2017 Jul;65(1):97-101. doi: 10.1097/MPG.0000000000001617. PMID 28471913

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 34 patients enrolled; 33 patients completed the study from 11 U.S. sites.
Pre-assignment Details: 33 eligible patients according to the inclusion/exclusion criteria were randomized in Period B (double-blind crossover) to the study.
Groups:
- Period A: Clinical Treatment Practice (Days -7 to -1): Period A was a 7-day baseline period. Patients received Peptamen 1.5 at their normal volume of enteral formula administration up to a maximum of 1000 mL per feeding. Current treatment practice was followed with normal use of oral pancreatic enzyme replacement therapy (PERT) during daily meals and nightly enteral feedings. A gastrointestinal symptom diary was completed for 7 consecutive days. Baseline Day -7 required a clinic visit followed by Days -6 to -1 at home.
- Crossover Period B: Placebo Then RELiZORB: Eligible subjects were randomized to Placebo then RELiZORB.
- Crossover Period B: RELiZORB Then Placebo: Eligible subjects were randomized to RELiZORB then Placebo.
- Period C: Clinical Treatment Practice + RELiZORB (Days 12-20): Period C was the open label clinical treatment period with RELiZORB. All patients used RELiZORB with Impact Peptide 1.5 at their normal volume as in Period A up to a maximum of 1000 mL per feeding. Patients were instructed to use the same daily dose and schedule of oral PERT taken in Period C as in Period A. There were no dietary restrictions. A gastrointestinal symptom diary was completed for 7 consecutive days. Patients received enteral feeding at home from Days 12 to 18 and returned to clinic for their end of study Day 19.
Period: Period A: Days -7 to -1
Arm/Group | Period A: Clinical Treatment Practice (Days -7 to -1) | Crossover Period B: Placebo Then RELiZORB | Crossover Period B: RELiZORB Then Placebo | Period C: Clinical Treatment Practice + RELiZORB (Days 12-20)
Started | 34 | 0 | 0 | 0
Completed | 33 | 0 | 0 | 0
Not Completed | 1 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0
Period: Period B: Days 1 to 11
Arm/Group | Period A: Clinical Treatment Practice (Days -7 to -1) | Crossover Period B: Placebo Then RELiZORB | Crossover Period B: RELiZORB Then Placebo | Period C: Clinical Treatment Practice + RELiZORB (Days 12-20)
Started | 0 | 17 | 16 | 0
Completed | 0 | 17 | 16 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Period C: Days 12 to 20
Arm/Group | Period A: Clinical Treatment Practice (Days -7 to -1) | Crossover Period B: Placebo Then RELiZORB | Crossover Period B: RELiZORB Then Placebo | Period C: Clinical Treatment Practice + RELiZORB (Days 12-20)
Started | 0 | 0 | 0 | 33
Completed | 0 | 0 | 0 | 33
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population
Groups:
- Clinical Treatment Practice: Period A: Days -7 to -1: Period A was a 7-day baseline period. Patients received Peptamen 1.5 at their normal volume of enteral formula administration up to a maximum of 1000 mL per feeding. Current treatment practice was followed with normal use of oral pancreatic enzyme replacement therapy (PERT) during daily meals and nightly enteral feedings. A gastrointestinal symptom diary was completed for 7 consecutive days. Baseline Day -7 required a clinic visit followed by Days -6 to -1 at home.
Arm/Group | Clinical Treatment Practice: Period A: Days -7 to -1
Number analyzed (Participants) | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 27
  Between 18 and 65 years | 6
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 28
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 31
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants] — 11 United States clinical sites.
  Participants
    United States | 33
Baseline Weight [Mean (Standard Deviation); unit: kilograms] — Population: Baseline weight obtained in Period A.
  kilograms | 41.81 (13.332)
Baseline Height [Mean (Standard Deviation); unit: centimeters] — Safety Population: Baseline Height Population: Baseline height obtained in Period A.
  centimeters | 152.32 (19.640)
Baseline Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] — Population: Baseline Body Mass Index obtained in Period A.
  kg/m^2 | 17.47 (2.026)

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Adverse Events and Unanticipated Adverse Device Effects
Description: 1) Frequency and severity of adverse events; 2) Patients with at least one unanticipated adverse device effects (UADE)
Time Frame: 27 days
Population: Safety Population
Measure: Count of Participants; unit: Participants
Groups:
- Crossover Period B: Placebo; Crossover Period B: RELiZORB: Non-gastrointestinal adverse events during administration.
- Clinical Treatment Practice + RELiZORB: Period C: Days 12-20: Non-gastrointestinal adverse events during CTP+RELiZORB administration.
Arm/Group | Clinical Treatment Practice: Period A: Days -7 to -1 | Crossover Period B: Placebo | Crossover Period B: RELiZORB | Clinical Treatment Practice + RELiZORB: Period C: Days 12-20
Number analyzed (Participants) | 33 | 33 | 33 | 33
Participants
  Patients With Adverse Events | 4 | 6 | 1 | 2
  Adverse Event by Severity (Mild) | 2 | 6 | 1 | 0
  Adverse Event by Severity (Moderate) | 2 | 0 | 0 | 1
  Adverse Event by Severity (Severe) | 0 | 0 | 0 | 1
  Patients With At Least One UADE | 0 | 0 | 0 | 0

2. Primary Outcome: Long Chain Polyunsaturated Fatty Acid Plasma Concentration (Intent to Treat Population)
Description: AUC analysis of plasma fatty acid concentration for DHA + EPA baseline adjusted over 24-hours
Time Frame: Day 1 first intervention and Day 9 second intervention.
Measure: Mean (Standard Deviation); unit: ug*h/mL
Groups:
- RELiZORB: Subjects receiving RELiZORB at any time in the study.
- Control: Subjects receiving placebo at any time in the study.
Arm/Group | RELiZORB | Control
Number analyzed (Participants) | 33 | 33
ug*h/mL | 536.98 (400.519) | 192.18 (198.664)
Statistical Analysis 1: Comparison: RELiZORB vs Control; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; The independent variables in the mixed model analysis included fixed effect factors for treatment (placebo or RELiZORB)

3. Other Pre Specified Outcome: Ease of Use of RELiZORB (Per-Protocol Population)
Description: Effect of enteral nutrition on select activities of daily living. Patients judged the size of breakfast after overnight enteral tube feeding with the following choices: No breakfast; Small breakfast; Normal breakfast; Big breakfast; Other.
Time Frame: Period C: Single assessment on Day 19 or 20
Population: Per Protocol Population.
Measure: Count of Participants; unit: Participants
Groups:
- Clinical Treatment Practice and Relizorb: Period C: Days 12-20: Period C was the open label clinical treatment period with RELiZORB. All patients received RELiZORB with Impact Peptide 1.5 at their normal volume as in Period A up to a maximum of 1000 mL per feeding. Patients were instructed to use the same daily dose and schedule of oral PERT taken in Period C as in Period A. There were no dietary restrictions. A gastrointestinal symptom diary was completed for 7 consecutive days. Patients received enteral feeding at home from Days 12 to 18 and returned to clinic for their end of study Day 19.
Arm/Group | Clinical Treatment Practice and Relizorb: Period C: Days 12-20
Number analyzed (Participants) | 32
Participants
  No breakfast | 11
  Small breakfast | 14
  Normal breakfast | 6
  Big breakfast | 0
  Other | 1

ADVERSE EVENTS:
Time Frame: 20 days
Description: Safety Population: Non-gastrointestinal Adverse Event by System Organ Class and Preferred Term (n=33)
Groups:
- Double-Blind Crossover: Period B: Days 1 to 11: Period B was the randomized, double-blind, placebo-controlled crossover period. Eligible patients were randomized in a 1:1 ratio to either Placebo-RELiZORB or RELiZORB-Placebo treatment sequences. On two separate administration Days 1 and 9, patients received 500 mL of Impact Peptide1.5 in clinic over a 4h period. Motility and acid suppression medications were discontinued 24h before arrival in clinic. No nocturnal feeding occurred between Days 1-2 and Days 9-10. During the home washout period Days 2 to 8, patients received Peptamen 1.5 for enteral nutrition up to a maximum volume of 1000 mL per feeding. Safety follow up calls were conducted on Days 2 and 10.
Arm/Group | Clinical Treatment Practice: Period A: Days -7 to -1 | Double-Blind Crossover: Period B: Days 1 to 11 | Clinical Treatment Practice and Relizorb: Period C: Days 12-20
Serious Adverse Events (participants affected / at risk) | 1/33 | 0/33 | 0/33
Other Adverse Events (participants affected / at risk) | 2/33 | 0/33 | 0/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clinical Treatment Practice: Period A: Days -7 to -1 (N=33) | Double-Blind Crossover: Period B: Days 1 to 11 (N=33) | Clinical Treatment Practice and Relizorb: Period C: Days 12-20 (N=33)
Cystic fibrosis pulmonary exacerbation (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) — Cystic fibrosis (increased cough, vomiting, decreased PFTs, hospital care required supplemental oxygen, IV antibiotics, and supportive care).
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clinical Treatment Practice: Period A: Days -7 to -1 (N=33) | Double-Blind Crossover: Period B: Days 1 to 11 (N=33) | Clinical Treatment Practice and Relizorb: Period C: Days 12-20 (N=33)
Headache (Nervous system disorders) | 2 (3) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less